CLINICAL TRIAL: NCT05072444
Title: A Phase 1, Randomized, Double-Blind, Single-Dose, Drug-Drug Interaction Study to Determine the Impact of Co-administration of QPX7728 on the Pharmacokinetics of QPX2014 in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study of IV QPX2014 Combined With QPX7728 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Qpex-201
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-02

CONDITIONS: Bacterial Infections
Keywords: beta-lactam antibiotic
MeSH Terms: conditions — Bacterial Infections | interventions — QPX7728

STUDY DESIGN:
Intervention Model Description: Double-Blind, Single-Dose, Drug-Drug Interaction Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind, Single-Dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- QPX7728 (Experimental): Drug: QPX7728 beta lactamase inhibitor Other names: IV
  Interventions: Drug: QPX7728; Drug: QPX2014
- QPX2014 (Experimental): Drug: QPX2014 antibiotic Other names: IV
  Interventions: Drug: QPX2014

INTERVENTIONS:
Drug: QPX7728 — beta lactamase inhibitor
  Other Names: IV
  Arms: QPX7728
Drug: QPX2014 — antibiotic
  Other Names: IV

SUMMARY:
QPX7728 is an ultra-broad-spectrum beta-lactamase inhibitor, with activity against numerous beta-lactamases, including class A extended spectrum betalactamases (ESBLs), class C cephalosporinases, and extended spectrum class D oxacillinases (OXA) that can hydrolyze cephalosporins and can be found in Enterobacteriaceae and Pseudomonas aeruginosa (P. aeruginosa). QPX7728 is also a potent inhibitor of carbapenemases from all molecular classes, such as class A Klebsiella pheumoniae carbapenemase (KPC), class B New-Dehli Metalo-beta-lactamase (NDM) and Verona integron-encoded metallo-betalactamase (VIM), and class D OXA-48 that are found in carbapenem resistant Enterobacteriaceae, and also class D carbapenemases such as OXA-23 that are found in carbapenem resistant Acinetobacter baumannii.

DETAILED DESCRIPTION:
The Centers for Disease Control (CDC) has listed carbapenem-resistant Enterobacteriaceae and Acinetobacter as urgent threats and multidrug resistant Pseudomonas, and extended spectrum beta-lactamase (ESBL)-producing Enterobacteriaceae as serious threats [CDC, 2019]. Consistent with the global nature of these resistant bacteria, the World Health Organization (WHO) has designated carbapenem-resistant, ESBL-producing Enterobacteriaceae, carbapenem-resistant Acinetobacter baumannii, and carbapenem-resistant Pseudomonas aeruginosa as pathogens for which new agents are critically needed [WHO, 2017]. Qpex Biopharma is developing a fixed combination antibiotic of QPX2014 plus an ultra-broad spectrum beta-lactamase inhibitor, QPX7728.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females of non-childbearing potential, 18 to 55 years of age (inclusive) at the time of screening.
2. Body mass index (BMI) ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive) at the time of screening.
3. Medically healthy with clinically insignificant screening results (e.g., laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination) as assessed by the PI.
4. Voluntarily consent to participate in the study.
5. Male volunteers must agree to be sexually abstinent or agree to use a condom when engaging in any sexual activity from study check-in (on Day -1) through 30 days following the last administration of the study drug, and to not donate sperm during this same period of time. If engaging in sexual activity with a female partner of childbearing potential, an additional method of birth control must be used.

   Approved additional methods of birth control include:
   1. Intrauterine device (IUD) in place for at least 3 months prior to Day 1 through 30 days following the final dosing of the study drug.
   2. Barrier method (diaphragm) for at least 14 days prior to Day 1 through 30 days following dosing of the study drug.
   3. Stable hormonal contraceptive for at least 3 months prior to Day 1 through 30 days following dosing of the study drug.
   4. Surgical sterilization (vasectomy) at least 6 months prior to Day 1.
6. Females of non-childbearing potential must be either postmenopausal (defined as 12 months spontaneous amenorrhea) with a serum FSH ≥ 40 mIU/mL or have undergone one of the following sterilization procedures at least 6 months prior to Day 1 (and is documented):

   1. Bilateral tubal ligation;
   2. Hysterectomy;
   3. Hysterectomy with unilateral or bilateral oophorectomy;
   4. Bilateral oophorectomy.

Exclusion Criteria:

1. History or presence of significant (based on the PI assessment) cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
2. Positive pregnancy test at screening or check-in (Day 1) for women.
3. Positive urine drug/alcohol testing at screening or check-in (Day -1). A repeat test may be performed at the Investigator's discretion in circumstances where a positive result is suspected to be caused by consumption of non-illicit substances.
4. Positive pregnancy test at screening or check-in (Day 1) for women.
5. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
6. History or presence of alcoholism or drug abuse within the 2 years prior to Day 1.
7. Use of more than an average of 5 packs/week of tobacco/nicotine-containing product within 6 months prior to Day 1. Subjects must agree to refrain from smoking within 48 hours prior to confinement and for the duration of the study.
8. Excessive intake of alcohol, defined as an average daily intake of greater than 2 standard drinks for women and 4 standard drinks for men, (1 bottle of beer (375mL) is equivalent to approximately 1.4 standard drinks, 1 glass of spirits (30mL) is equivalent to approximately 1 standard drink and 1 glass (150mL) of wine is equivalent to approximately 1.5 standard drinks).
9. Use of any prescription medication (with the exception of hormone replacement therapy for females) within 14 days prior to Day 1.
10. Use of any over-the-counter (OTC) medication, including herbal products, probiotics and vitamins, within the 7 days prior to Day 1. Up to 2 grams per day of acetaminophen is allowed for acute events at the discretion of the PI.
11. Use of antacids, H2 receptor blockers or proton pump inhibitors within 3 days prior to Day 1.
12. Documented hypersensitivity reaction or anaphylaxis to any medication, including beta-lactam antibiotics.
13. Blood donation or significant blood loss (i.e., > 500 mL) within 56 days prior to Day 1.
14. Plasma donation within 7 days prior to Day 1.
15. Participation in another investigational clinical trial within 30 days prior to Day 1 or within 5 half-lives of the previous investigational drug, whichever is longer.
16. Surgery within the past three months prior to Day 1 determined by the PI to be clinically relevant. Minor surgeries allowed include laser vision, minor dental and tooth extraction, mole or basal cell skin removal, endoscopy, and biopsy.
17. Any significant acute illness (based on the PI assessment) within 30 days prior to Day 1.
18. QTcF interval >450 msec for males and >470 msec for females or history of prolonged QT syndrome at screening or check-in (Day -1).
19. Calculated creatinine clearance less than 80 mL/min (Cockcroft- Gault method) at screening or check-in (Day -1).
20. Subjects who have any clinically significant laboratory value abnormalities at screening or check-in (Day -1), in particular:

    1. White blood cell count < 3,000/mm3, hemoglobin < 11g/dL.
    2. Absolute neutrophil count < 1,200/mm3 or platelet count < 120,000/mm3.
21. Liver function abnormalities at screening or check-in (Day -1) (defined by an elevation in bilirubin, AST or ALT > ULN for subjects based on age and sex).
22. Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study.
23. Participation in a previous QPX7728 or QPX7831 study.
24. Participation of research site staff, their close family, or significant others.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) between dosing groups | up to 9 days
  Comparison will be performed between the dosing groups for AUC. Mean graphical presentation of the data will be reported.
  Statistical analysis of exposure parameters will be performed.
Peak plasma Concentration measurements by subject and by dosing group | up to 9 days
  Comparison will be performed between the dosing groups. Mean graphical presentation of the data will be reported.
  Statistical analysis of exposure parameters will be performed.
Urine Pharmacokinetic (PK) amount excreted by subject and by dosing group | up to 9 days
  Urine PK parameters such as amount excreted will be calculated from urinary excretion data
Urine PK % dose excreted by subject and by dosing group | up to 9 days
  Urine PK parameters such as amount of % dose excreted will be calculated from urinary excretion data
Incidence of Treatment -Emergent Adverse events (AEs) by subject and by dosing group | up to 9 days
  Number of patients with Treatment-Emergent AEs by treatment arm, severity and relationship to treatment
Number of patients with changes from baseline in safety parameters | up to 9 days
  Number of patients with changes in safety parameters before and after dosing by subject and treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S Loutit, MBChB, Study Director — Qpex Biopharma, Inc.
Locations (1):
- Altasciences, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No